CLINICAL TRIAL: NCT02119728
Title: A Randomized Multicenter Phase II Study Using HPPH With PDT Versus Standard of Care Surgery for Patients With T1/T2 Squamous Cell Carcinoma of the Oral Cavity
Brief Title: Photodynamic Therapy With HPPH in Treating Patients With Squamous Cell Carcinoma of the Oral Cavity
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 246513; NCI-2014-00756 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 246513 (Other: Roswell Park Cancer Institute); P01CA055791 (NIH); P30CA016056 (NIH)
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage I Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage I Squamous Cell Carcinoma of the Oropharynx; Stage I Verrucous Carcinoma of the Oral Cavity; Stage II Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage II Squamous Cell Carcinoma of the Oropharynx; Stage II Verrucous Carcinoma of the Oral Cavity; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Verrucous Carcinoma of the Oral Cavity
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (standard of care surgery) (Active Comparator): Patients undergo standard of care surgery on day 1.
  Interventions: Procedure: therapeutic conventional surgery
- Arm II (HPPH, photodynamic therapy) (Experimental): Patients receive HPPH IV over 1 hour on day 0. Approximately 24 hours later, patients undergo photodynamic therapy on day 1.
  Interventions: Drug: HPPH; Device: Light Infusion Therapy™

INTERVENTIONS:
Drug: HPPH — Undergo photodynamic therapy with HPPH
  Other Names: Photochlor
  Arms: Arm II (HPPH, photodynamic therapy)
Device: Light Infusion Therapy™ — Undergo photodynamic therapy with HPPH
  Other Names: PDT; therapy, photodynamic
  Arms: Arm II (HPPH, photodynamic therapy)
Procedure: therapeutic conventional surgery — Undergo standard of care surgery
  Arms: Arm I (standard of care surgery)

SUMMARY:
This randomized phase II trial studies how well photodynamic therapy with HPPH works in treating patients with squamous cell carcinoma of the oral cavity. Photodynamic therapy uses HPPH that becomes active when it is exposed to a certain kind of light. When the drug is active, cancer cells are killed. This may be effective against squamous cell carcinoma of the oral cavity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the non-inferiority of photodynamic therapy (PDT) to standard of care surgery.

SECONDARY OBJECTIVES:

I. To determine improvement in quality of life (QoL) using the University of Washington Quality of life questionnaire version 4.

II. To assess the toxicity using the Cancer Therapy Evaluation Program (CTEP) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 4.0).

III. To explore progression-free survival in this patient population treated with HPPH mediated PDT.

TERTIARY OBJECTIVES:

I. Immune markers (T cells). II. To investigate the correlation of the tri-modal optical spectroscopy with tumor response to PDT.

OUTLINE: Patients are randomized to 1 of 2 treatments arms.

ARM I: Patients undergo standard of care surgery on day 1.

ARM II: Patients receive HPPH intravenously (IV) over 1 hour on day 0. Approximately 24 hours later, patients undergo photodynamic therapy on day 1.

After completion of study treatment, patients are followed up 3-4 months for 1 year, 3-6 months for 1 year, 4-8 months for 1 year, and once a year for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patients with Tl/T2 squamous cell carcinoma of the oral cavity with or without extension to the oropharynx
* Histologically confirmed squamous cell carcinoma of the target tumor(s)
* Tumor thickness is 4 mm or less (in the judgment of the physician)
* Computed tomography (CT) of the neck to confirm staging
* Tumor accessible for unrestricted illumination for photodynamic therapy (PDT) (accessibility as determined by the physician)
* Life expectancy of at least 12 months in the judgment of the physician
* Patients of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Patient or legal representative must understand the investigational nature of this study and sign an Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy or targeted agents within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients with known brain metastases should be excluded from this clinical trial
* Patients with porphyria, or with known hypersensitivity to porphyrins or porphyrin-like compounds
* White blood cells (WBC) < 4,000
* Total serum bilirubin > 2 mg/dL
* Serum creatinine > 2 mg/dL
* Alkaline phosphatase (hepatic) > 3 times the upper normal limit
* Serum glutamic oxaloacetic transaminase (SGOT) > 3 times the upper normal limit
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Nodal disease as detected by clinical exam or CT
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive study drug
* Received an investigational agent within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Objective tumor response assessed according to Response Evaluation Criteria in Solid Tumors version 1.1 | 3 months after treatment
  Objective tumor response will be tabulated overall. Tumor response will be determined by comparing photographs of the treated site (with reference ruler) before and after PDT. Efficacy (e.g., tumor response) will be estimated using simple relative frequencies. The corresponding 95% confidence intervals for the estimated probabilities will be computed using the method proposed in Clopper and Pearson.
Changes in quality of life evaluated by the University of Washington Quality of Life Questionnaire version 4 | Baseline to up to 5 years
  In the analysis of QoL simple data analyses will initially take place including individual patient level profile plots and overall mean plots used to examining the mean structure. Formal statistical examination of longitudinal patterns will be done through the use of a mixed model. All tests will be two-sided and tested at a 0.05 nominal significance level. Standard diagnostic plots will be used to assess model fit and transformations of variables may be considered in order to meet statistical assumptions.

SECONDARY OUTCOMES:
Frequency of toxicity graded according to NCI CTCAE version 4.0 | Up to 6 weeks after treatment
  The frequency of toxicities will be tabulated by grade across all cycles. The safety of the interventions will be assessed through the evaluation of grade 3 or higher toxicities deemed possibly related to treatment. Toxicity rates will be estimated using simple relative frequencies. The corresponding 95% confidence intervals for the estimated probabilities will be computed using the method proposed in Clopper and Pearson.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Arshad, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States